CLINICAL TRIAL: NCT06664606
Title: Satisfaction and Knowledge Acquisition Following a Pain Neuroscience Education Program in Primary Students with and Without Intellectual Disabilities
Brief Title: Impact of a Pain Neuroscience Education Program on Primary Students with and Without Intellectual Disabilities
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, Clinical Professor, Universidad de Extremadura
Other Study IDs: 06
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pain (back / Neck)
Keywords: Pain Management; Health Education; Students; Neuroscience
MeSH Terms: conditions — Chronic Pain; Agnosia; Health Education

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Students in Rural Public Schools: This group consists of primary school students from rural public schools in Extremadura, Spain, participating in a Pain Neuroscience Education (PNE) program.
  Interventions: Behavioral: Pain Neuroscience Education Program (PNE)
- Students in Urban Public Schools: This group includes primary school students from urban public schools in Extremadura, Spain, who participated in a Pain Neuroscience Education (PNE) program.
  Interventions: Behavioral: Pain Neuroscience Education Program (PNE)
- Students in Special Education Schools: This group consists of students from special education schools in Extremadura, Spain, who have intellectual disabilities. These students participated in the Pain Neuroscience Education (PNE) program, with the goal of understanding program effectiveness in an inclusive educational environment tailored to students with intellectual disabilities.
  Interventions: Behavioral: Pain Neuroscience Education Program (PNE)
- Students in Regular Education Schools: This cohort includes primary school students from regular education schools in Extremadura, Spain, without intellectual disabilities. These students participated in the Pain Neuroscience Education (PNE) program, providing insights into the program's impact on general education settings and comparing outcomes with other cohorts.
  Interventions: Behavioral: Pain Neuroscience Education Program (PNE)

INTERVENTIONS:
Behavioral: Pain Neuroscience Education Program (PNE) — The Pain Neuroscience Education (PNE) Program is a structured educational intervention aimed at primary school students with and without intellectual disabilities. This program introduces students to basic concepts of pain neuroscience, designed to increase understanding of pain mechanisms and promote healthy pain coping strategies. The intervention was adapted to 'easy reading' format to ensure accessibility for students with intellectual disabilities, and was delivered in both rural and urban school settings in Extremadura, Spain.

SUMMARY:
This observational study evaluates the impact of a Pain Neuroscience Education (PNE) program on primary school students in Extremadura, Spain. The study examines satisfaction levels and knowledge acquisition regarding pain neuroscience among students with and without intellectual disabilities. Conducted across both rural and urban educational centers, as well as special and regular education schools, this study aims to identify the effectiveness of PNE in enhancing pain-related knowledge and addressing Sustainable Development Goals (SDGs) awareness. Additionally, the program includes interactive educational activities tailored for accessibility, using resources such as easy-to-read questionnaires and hands-on models, to support inclusive health education. Data collection involves pre- and post-intervention questionnaires to assess satisfaction and knowledge gains, with statistical analysis exploring differences between demographic and school-type groups.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the fifth or sixth grade of primary education in schools within the Autonomous Community of Extremadura.
* Students who regularly attend academic activities and complete the educational intervention.

Exclusion Criteria:

* Students who do not attend school regularly or who are not expected to complete the intervention.
* Students with severe cognitive or behavioral impairments that may interfere with participation in the educational activities.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of fifth and sixth grade primary school students enrolled in the Autonomous Community of Extremadura, Spain. The participants include students from both regular and special education schools, encompassing both urban and rural areas. The sample represents a diverse group with variations in intellectual abilities, aiming to assess the impact of a neuroscience education program on understanding pain and promoting health knowledge.
Sampling Method: Non-Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Satisfaction Level and Knowledge Acquisition in Pain Neuroscience Education | Immediately after completion of the educational intervention
  This study measures the level of satisfaction and the knowledge acquired by primary school students with and without intellectual disabilities following participation in a Pain Neuroscience Education (PNE) program. Satisfaction and knowledge are assessed through a structured questionnaire, focusing on three main dimensions: training activity, teacher's role, and understanding of Sustainable Development Goals (SDGs) related to health. The responses are analyzed to evaluate the program's impact across different educational settings, including rural vs. urban and special vs. regular education

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo-Antúnez, Ph.D., Study Director — University of Extremadura
Locations (1):
- Universidad de Extremadura, Badajoz, Badajoz, Spain